CLINICAL TRIAL: NCT02007122
Title: Multiple-dose Pharmacokinetics of Ceftaroline During Continuous and Intermittent Renal Replacement Therapy in Patients Requiring Renal Replacement Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, Univ.-Prof. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEFTAROLINE_RRT
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Infection During Renal Replacement Therapy
Keywords: HD; CVVH; renal replacement therapy; ceftaroline; pharmacokinetics
MeSH Terms: interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IRRT (Experimental): Ceftaroline levels are measured in patients receiving intermittent renal replacement therapy
  Interventions: Other: Ceftaroline in IRRT
- CRRT (Experimental): Ceftaroline levels are measured in patients receiving continuous renal replacement therapy
  Interventions: Other: Ceftaroline in CRRT

INTERVENTIONS:
Other: Ceftaroline in CRRT — Plasma levels of ceftaroline will be measured in patients receiving CRRT
  Arms: CRRT
Other: Ceftaroline in IRRT — Ceftaroline plasma levels will be measured in patients receiving intermittent renal replacement therapy
  Arms: IRRT

SUMMARY:
The study will be conducted to investigate the pharmacokinetics of ceftaroline during continuous and intermittent renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, able to give written informed consent
* Suspected or proven bacterial infection requiring parenteral antibiotic therapy.
* Renal replacement therapy (continuous or intermittent)

Exclusion Criteria:

* Known hypersensitivity to ceftaroline or other cephalosporins, or severe hypersensitivity (anaphylactic reaction) to beta-lactam antibacterial agents.
* An expected survival of less than two days.
* Known pregnancy
* Coadministration of valproic acid or probenecid, which cannot be discontinued for the duration of the study
* Ceftaroline as monotherapy for resistent species or fungal infections.
* Other reasons oposing the study participation on the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Influence of renal replacement therapy on the area under concentration curve of ceftaroline plasma concentration levels. | day 15
  Pharmacokinetic samples are drawn on multiple timepoints from each patient during his participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria